CLINICAL TRIAL: NCT02492620
Title: A Two-Arm, Open-Label, Standard of Care Control Evaluation of Ferric Citrate for the Transition From Chronic Kidney Disease Stage 4/5 to Chronic Kidney Stage 5D
Brief Title: Ferric Citrate for the Transition From CKD Stage 4/5 to CKD Stage 5D
Acronym: 05D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05D
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia; Iron Deficiency Anemia; Renal Insufficiency
Keywords: ferric citrate; phosphate; kidney
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia; Anemia, Iron-Deficiency; Renal Insufficiency | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric Citrate (Active Comparator): Ferric citrate (FC) will be supplied as tablets containing 210mg of ferric iron (as 1g ferric citrate) to those subjects randomized to FC. These participants will be initiated on study drug with a fixed dose of FC beginning with 2 tablet per meal.
  Interventions: Drug: Ferric Citrate
- Standard of Care (SOC) (No Intervention): Participants may receive open-label, non-FC phosphate binders at the discretion of their treating physician. During the Dialysis Period, dose of phosphate binders, use of ESA, intravenous iron and blood transfusions will be at the discretion of the primary treating nephrologist. Participants assigned to the SOC treatment arm may not receive FC at any point during the study.

INTERVENTIONS:
Drug: Ferric Citrate — Auryxia (ferric citrate) is a non calcium based phosphate binder indicated for the control of serum phosphorus levels in patients with chronic kidney disease on dialysis
  Other Names: Auryxia
  Arms: Ferric Citrate

SUMMARY:
It is the investigators hypothesis that participants treated with Ferric Citrate (FC) during the non-dialysis CKD stage (4/5) with sufficient duration prior to initiating RRT, will result in improved biochemical control of anemia (Hb, TSAT) and mineral metabolism (P, FGF23) and furthermore, will result in a reduced need for ESA and intravenous iron. The investigators further hypothesize that effective treatment of anemia and mineral metabolism with FC in the pre-dialysis and transition period will result in improved physical functioning, reduced hospitalization and reduced total cost of care when compared to participants receiving contemporaneously provided standard of care therapy.

DETAILED DESCRIPTION:
This is an up to 50 week, phase 3, clinical trial in patients with estimated glomerular filtration rate (eGFR) ≤ 20 ml/min/1.73m2. It will be comprised of an up to 36-week non-dialysis period (NDP), or until such time as subjects require renal replacement therapy (RRT) with dialysis when they will immediately roll into a 12-week dialysis period (DP). The study will consist of up to 16 clinic visits over a maximum period of 50 weeks. There will be a screening period of up to 14 days after which subjects will be randomized into the NDP in a 2:1 ratio to receive either FC (n=150) or SOC (n=75). Each eligible participant will be randomized to either fixed dose open-label ferric citrate (FC) or standard of care (SOC) treatment. Participants randomized to SOC will receive care directed by their primary nephrologist throughout the study duration with the only restriction being that they cannot receive treatment with FC during the NDP or DP. Participants randomized to FC will receive it throughout the study duration.

220 participants were screened to randomize 200 subjects 2:1 (FC:SOC) into the NDP. It is anticipated that 35-45% of participants will reach the dialysis period (DP) during the 36 week follow up. Participants who initiate RRT with dialysis will enter the Dialysis Period (DP) during which those participants previously assigned to ferric citrate will continue to receive open-label ferric citrate and those previously assigned to SOC will receive open-label, non-FC phosphate binders at the discretion of their treating physician. During this period all participants will be treated to standard of care guidelines which suggest that if serum phosphate is above the upper limit of normal (4.5 mg/dL), it should be reduced. During the DP, dose of P binders, use of ESA, intravenous iron and blood transfusions will be at the discretion of the primary treating nephrologist. Participants assigned to the SOC treatment arm may not receive FC at any point during the study.

Only participants that begin permanent RRT with dialysis will be eligible to enter the 12 week DP. Participants that do not begin RRT after 9 months participation in the NDP will be deemed to have reach the end of study and have end of study procedures performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years at screening visit
2. Serum phosphate > or equal to 3.0 mg/dL obtained at screening
3. CKD with eGFR < or equal to 20 mL/min obtained at screening*
4. Hemoglobin (Hgb) >8.0 g/dL obtained at screening
5. TSAT <55% obtained at screening
6. Females of child bearing potential with negative serum pregnancy test obtained at screening
7. Willing and able to give written informed consent
8. Anticipated to have > or equal to 8 weeks prior to need for initiating RRT in the opinion of the investigator

Exclusion Criteria:

1. Liver enzymes (ALT/AST) >X3 times upper limit of normal at screening
2. Use of IV iron, blood transfusions or ESA agents within 2 weeks prior to the screening visit and prior to the Day 1 visit.
3. Evidence of acute kidney injury (i.e., no CKD) or planned need for RRT within 12 weeks of screening
4. Scheduled kidney transplant within 24 weeks of screening
5. Contra-indication to ferric citrate: iron overload syndrome, allergic reaction or known intolerance to ferric citrate
6. Clinically significant medical condition felt to interfere with tolerance of oral medication
7. Life expectancy < 6 months or confirmed conviction that subject does NOT want to initiate RRT despite a decline in kidney function
8. Active drug or alcohol dependence or abuse (excluding tobacco use or marijuana use) within the 12 months prior to screening (in the opinion of the PI)
9. Psychiatric disorder that interferes with the subject's ability to comply with the study protocol in the opinion of the PI
10. Any other medical condition that, in the opinion of the PI, renders the subject unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the subject
11. Inability to cooperate with study personnel or study procedures
12. Females who are pregnant or breastfeeding
13. Receiving or has received any investigational drug with in the past 30 days prior to the Day 1 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Serum phosphate value prior to starting renal replacement therapy | baseline

SECONDARY OUTCOMES:
Serum hemoglobin prior to starting renal replacement therapy | baseline
Serum transferrin saturation prior to starting renal replacement therapy | baseline
Serum fibroblast growth factor 23 prior to starting renal replacement therapy | baseline

OTHER OUTCOMES:
Cumulative dose of erythropoietin analog | Baseline visit to 90 days after starting renal replacement therapy
  Total dose of ESA received in units from baseline visit to 90 days post renal replacement
Cumulative dose of intravenous iron | Baseline visit to 90 days after starting renal replacement therapy
  Total dose of intravenous iron received in units from baseline visit to 90 days post renal replacement

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, P.C.
Locations (1):
- Denver Nephrologists, P.C., Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086